CLINICAL TRIAL: NCT00468065
Title: VeinViewer Assisted Intravenous Catheter Placement in the Pediatric Emergency Department
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lifespan (Other)
Responsible Party: Bruce Becker, Lifespan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0037-07
Record Dates: First submitted 2007-04-27; First posted 2007-05-01 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2007-04

CONDITIONS: Catheterization
Keywords: intravenous; catheter; IV

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): TO use Veinviewer to improve the effectiveness of IV starts in children
  Interventions: Device: VeinViewer
- B (No Intervention): Standard approach to placing IV s in children

INTERVENTIONS:
Device: VeinViewer — Veinveiwer is used to view veins subQ
  Arms: A
Device: Veinviewer — near infrared light reveals veins subcutaneously
  Arms: A

SUMMARY:
The objective of this study is to evaluate the effectiveness of the VeinViewer® near infrared device to facilitate the placement of intravenous catheters in children who require intravenous cannulation in the pediatric emergency department. This clinical protocol is designed to determine whether using the VeinViewer increases the ease and efficiency of IV cannulation (as perceived by the operator), decreases the time to effective cannulation, decreases the number of sticks and extravasations, and decreases the child's and the parents perception of the pain of IV cannulation.

DETAILED DESCRIPTION:
Needle sticks are part of many standard treatments in the pediatric emergency department (ED) and are frequently a source of pain and anxiety for children. Intravenous catheters (IVs) have been shown to be among the leading causes of pain in hospitalized children 1 and venipucture is commonly seen as one of the most painful and frequently performed invasive procedures by nurses. 2 (Jacobson et al.) Children recording VAS pain scores in response to IV catheter placement in the Emergency Department rated the pain as 3.23/5.0 and their parent rated their children's pain as 3.4/5.0. 3 (Skarbek et al.) The placement of intravenous catheters would be more efficient and less stressful if the clinician had a clear roadmap or picture highlighting the location of the vein. The lack a clear visual guide to IV placement often leads to multiple painful attempts at catheter placement as well as delays urgent in treatment ( I.V. fluid and medication administration) and increased use of human resources. The current average number of catheter punctures needed in order to achieve successful catheter placement is 2.4 with a range of 1-14. 4 ( Larue, GD ) The VeinViewer by Luminetx™ allows the clinician to clearly see the child's accessible vasculature or the lack thereof in real time, directly on the surface of the skin. The clinician can be trained to operate the VeinViewer in minutes and use does not require any additional job or skills certification. The VeinViewer is free standing and hands-free allowing the clinician the freedom to use both hands to carry out the work of placing the catheter (unlike ultrasound which requires one hand to hold the probe and the other hand to place the catheter, unless two people are available and able to coordinate their work efforts thus doubling the resources necessary for I.V. placement. The VeinViewer is non-invasive and causes no tissue damage. There is no patient contact with the device and therefore no risk of infectious disease contamination with blood products. The VeinViewer uses near-infrared light to locate subcutaneous veins and project their location onto the surface of the skin thus creating a visible roadmap for I.V catheter placement. This protocol describes a prospective, randomized, study, evaluating the effectiveness of VeinViewer in increasing the ease of intravenous cannulation in children receiving intravenous cannulation in the pediatric emergency department. The investigators hypothesize that cannulation using VeinViewerâ will require fewer sticks and will result in fewer missed or repeated IV starts, fewer extravasating ("blown vein") IV placements, increased perceived ease of placement by the operator, and decreased pain associated with the IV placement as perceived by the child, the parent, and the operator.

2. Background Intravenous cannulation is a routine and common part of treatment for children receiving care in the Pediatric Emergency Department. Intravenous cannulation is painful and often challenging in children. Peripheral IV's are generally placed using visual and/or tactile cues. These may be minimal or deceptive in children who often have small peripheral veins and increased subcutaneous fat with opaque, elastic skin. Health care workers often struggle to place these IV's successfully making multiple sticks, infiltrating subcutaneous tissues, requiring extensive operator time, and, most importantly, causing the patient and the parent distress. A number of approaches have been tried, attempting to decrease the pain of these cannulations. Most of these involve the cutaneous application of lidocaine in an attempt to numb the skin and decrease the pain of the stick.

EMLA and more recently, LMX (lidocaine in liposomal delivery system) are effective topical agents but there is a 30 minute dwell time - inappropriate in the Emergency Medicine setting. A number of devices have been tested which decrease the barrier of the stratum corneum thus allowing the lidocaine to anesthetize the skin in 3-5 minutes. These include a hand held laser (effective but burns and pigments the skin), a small ultrasound (effective but bulky and difficult to use), and gas pressure driven powdered lidocaine (effective but not approved by the FDA yet for general sales and distribution). These devices depend on identifying the vein and then successfully cannulating the identified vein through the anestethized skin. Missed sticks force the operator to begin the anesthesia process all over again in a different site. This process is time consuming and ineffective in the ED setting.

Other centers have begun to employ ultrasound to identify the veins for peripheral cannulation to cannulate under indirect visualization. This process is difficult for small mobile pediatric veins and requires extensive operator training and practice. It also requires an extra set of operator hands when children, often less than cooperative, are involved. It is unclear that this approach will be effective in the Pediatric ED.

Vein Viewerâ is a hands off device that projects a map of the subcutaneous veins onto the surface of the skin. It allows the operator to insert the IV catheter under direct visualization. It can be used by one operator who can insert the catheter and restrain the child's arm while using the device. Direct visualization is accurate and decreases the blind sticks, missed "fishing expeditions", and extravasations of IV fluid and medication (often not benign) that can occur with IV cannulation, especially in children. Decreasing the number of sticks and the time to successful catheterization will decrease the child's and the parents perceived pain of the procedure and the operator time to effective catheterization thus increasing the efficiency of the operator and the ED in general, and speeding the initiation of therapy (IV hydration or medication). The Vein Viewer has no side effects and is visually interesting to children and parents. It has the potential to revolutionize the effectiveness and efficiency, of IV cannulation in the Pediatric Emergency Department and decrease substantially the child's and the parent's perceived pain from the procedure and fear of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be children between the ages of 8-17 who present to the pediatric emergency department and require intravenous cannulation as part of their regular care
* Both the child and the parent/guardian must be English-speaking
* Both the child and the parent/guardian must be comfortable with the experimental protocol as explained to them by the study investigator or a research assistant
* The parent/guardian must be able to understand and sign informed consent and a HIPAA form
* The child must provide assent
* The child must demonstrate understanding of the 100mm standard Visual Analog Scale

Exclusion Criteria:

Participants must not have:

* Need for an emergent IV

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2007-04; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Time to successful placement of IV by practitioner | one hour

CONTACTS AND LOCATIONS:
Overall Officials: Bruce M Becker, Principal Investigator — Lifespan
Locations (1):
- Hasbro Children's Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Chapman LL, Sullivan B, Pacheco AL, Draleau CP, Becker BM. VeinViewer-assisted Intravenous catheter placement in a pediatric emergency department. Acad Emerg Med. 2011 Sep;18(9):966-71. doi: 10.1111/j.1553-2712.2011.01155.x. Epub 2011 Aug 19. PMID 21854488